CLINICAL TRIAL: NCT06463639
Title: A Retrospective Cohort Study of FLT3 Turnaround Time in Acute Myeloid Leukemia (AML) Patients and the Clonal Evolution of FLT3 in Relapse/Refractory AML Patients in National Taiwan University Hospital
Brief Title: FLT3 Clonal Evolution in Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 202203013RSD
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; FLT3; Clonal evolution
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective cohort study aims to describe the current FLT3 testing landscape in Taiwan. It includes two patient groups: non-M3 primary AML patients with relapsed/refractory disease (R/R cohort) and newly diagnosed non-M3 primary AML patients (newly diagnosed cohort).

Primary objectives:

Estimate FLT3 testing turnaround time in clinical practice. Assess FLT3 clonal evolution in the R/R cohort.

Secondary objectives:

Determine FLT3 mutation prevalence. Describe karyotypes, co-mutations, and allelic ratios in both cohorts. Study European LeukemiaNet (ELN) risk in the newly diagnosed cohort. Evaluate the association of FLT3 mutation changes with treatment discontinuation and overall survival (OS) in the R/R cohort.

Investigate the link between Measurable Residual Disease (MRD) outcomes with treatment discontinuation and OS in the newly diagnosed cohort.

Data from the National Taiwan University Hospital integrated Medical Database (NTUH-iMD) and NTUH-AML dataset will be used. The index date is the earliest R/R AML evidence for the R/R cohort and the initial AML diagnosis date for the newly diagnosed cohort. A three-year baseline period will provide patient history and comorbidity information. Patients will be followed until the study's end, loss to follow-up, or death.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a heterogeneous group of hematological diseases. According to the Taiwan Cancer Registry Annual Report, 859 new AML cases were diagnosed in Taiwan in 2018, with an age-standardized incidence rate of 3.06 in males and 2.18 in females per 100,000 person-years.

The FMS-like tyrosine kinase 3 gene (FLT3) affects the proliferation and differentiation of stem cells or hematopoietic progenitor cells. FLT3 mutations are found in 25-30% of newly diagnosed AML patients and are considered a negative prognostic factor, remaining significant even after intensive chemotherapy and/or stem cell transplant.

Two critical issues for ensuring timely targeted therapy for FLT3+ patients are the speed of FLT3 test turnaround and the use of tests at key time points. Rapid turnaround times are necessary for early intervention, with European LeukemiaNet (ELN) recommending results within 3 days. However, it's unclear if this is achievable in real-world settings. FLT3 mutation status evolves, with 15-25% of patients losing and 13% acquiring the mutation at relapse. Despite guidelines recommending FLT3 testing at diagnosis and relapse, there is no consensus in Taiwan on its importance and timing.

Some observational studies on AML in Taiwan have been conducted but provide limited information on the timing and turnaround of FLT3 testing in real-world practice.

This study will describe the current FLT3 testing landscape, including turnaround time and timing of tests among adult relapsed/refractory (R/R) AML patients at NTUH. It will also investigate the clinical characteristics and survival outcomes of both adult R/R AML and newly diagnosed AML patients.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed/refractory cohort:

  1. Adult patient (age ≥18 years) diagnosed with non-M3 primary AML (confirmed diagnosis using WHO 2016 criteria within the NTUH-AML dataset) who:
  * First experienced refractory disease (failure to achieve complete remission or complete remission with incomplete hematologic recovery) to 2 cycles of induction therapy between 1 January 2009 and 31 December 2019, OR
  * First experienced hematological relapse after a CR between 1 January 2009 and 31 December 2019. Patient with bone marrow blasts ≥5 %, reappearance of blasts in the blood, or development of extramedullary disease after achieving remission is defined to have relapse of AML.
* Newly diagnosed cohort:

  1. Adult patient (age ≥ 18 years) newly diagnosed with non-M3 primary AML (confirmed diagnosis using WHO 2016 criteria within the NTUH-AML dataset) between 1 January 2009 and 31 December 2019.

Exclusion Criteria:

* Relapsed/refractory cohort:

  1. Patient with M3 subtype (acute promyelocytic leukemia, APL)
  2. Patient with prior history of myelodysplastic syndrome (MDS) or myeloproliferative neoplasms (MPN)
  3. Patient without any FLT3 records
  4. Patient with secondary or therapy-related AML
* Newly diagnosed cohort:

  1. Patient with M3 subtype (APL)
  2. Patient with prior history of MDS or MPN
  3. Patient without any FLT3 records
  4. Patient with secondary or therapy-related AML

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: FLT3 testing was introduced in NTUH since 2000 and became a standard test since 2015, while MRD testing became standard and widely used since 2009. Thus, eligible patients for the R/R cohort and the newly diagnosed cohort will be identified between the period of 1 January 2009 and 31 December 2019.
Sampling Method: Non-Probability Sample
Enrollment: 1213 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Estimate FLT3 testing turnaround time in clinical practice. | From date of diagnosis until the date of death from any cause, assessed up to 30 years
  This outcome measure focuses on determining the average time required to complete FLT3 testing from the point of sample collection to the delivery of results in a real-world clinical setting. The goal is to evaluate the efficiency and speed of the current FLT3 testing processes. By estimating the turnaround time, the investigators aim to identify potential delays and areas for improvement to ensure timely initiation of targeted therapies for patients with acute myeloid leukemia (AML). This data will provide valuable insights into the operational aspects of FLT3 testing and its alignment with clinical practice guidelines.
Assess FLT3 clonal evolution in the relapsed/refractory cohort. | From date of diagnosis until the date of death from any cause, assessed up to 30 years
  This outcome measure involves analyzing the changes in FLT3 mutation status in patients with relapsed or refractory acute myeloid leukemia (AML). The study aims to track the presence, loss, or acquisition of FLT3 mutations over the course of the disease. By examining FLT3 clonal evolution, the investigators aim to better understand how these genetic changes correlate with disease progression, treatment response, and overall patient outcomes. The results will provide insights into the dynamics of FLT3 mutations and inform future therapeutic strategies.

SECONDARY OUTCOMES:
Determine FLT3 mutation prevalence at diagnosis | From date of diagnosis until the date of death from any cause, assessed up to 30 years
  This outcome measure aims to establish the prevalence of FLT3 mutations in patients newly diagnosed with acute myeloid leukemia (AML). By identifying the proportion of patients who test positive for FLT3 mutations at the time of diagnosis, the investigators can better understand the genetic landscape of AML within the study population. This data is crucial for assessing the potential impact of FLT3-targeted therapies and for tailoring treatment strategies according to mutation status
Evaluate the association of FLT3 mutation changes with treatment discontinuation and overall survival (OS) in the relapsed/refractory cohort. | From date of diagnosis until the date of death from any cause, assessed up to 30 years
  This outcome measure investigates how changes in FLT3 mutation status (acquisition, loss, or maintenance) are associated with treatment discontinuation and overall survival (OS) in patients with relapsed or refractory acute myeloid leukemia (AML). By examining the relationship between FLT3 clonal evolution and clinical outcomes, the investigators aim to determine the prognostic significance of these genetic changes.
Investigate the link between Measurable Residual Disease (MRD) outcomes with treatment discontinuation and OS in the newly diagnosed cohort. | From date of diagnosis until the date of death from any cause, assessed up to 30 years
  This outcome measure examines the relationship between Measurable Residual Disease (MRD) status and key clinical outcomes, specifically treatment discontinuation and overall survival (OS), in patients newly diagnosed with acute myeloid leukemia (AML). By assessing MRD levels at various stages of treatment, the investigators aim to determine how residual disease impacts the likelihood of continuing therapy and the overall prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided